CLINICAL TRIAL: NCT07204041
Title: Efficacy and Safety of XTD Regimen (Selinexor, Thalidomide and Dexamethasone) in Adult Patients With Relapsed/Refractory Langerhans Cell Histiocytosis: A Prospective, Multicenter, Single-Arm Study.
Brief Title: Efficacy and Safety of XTD Regimen (Selinexor, Thalidomide and Dexamethasone) in Adult Patients With Relapsed/Refractory LCH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH0027
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Langerhans Cell Histiocytosis (LCH)
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — selinexor; Thalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, interventional study, with a planned number of subjects: approximately 40 cases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with relapsed or refractory LCH (Experimental): (1) Relapsed or refractory LCH; (2) Age ≥ 18 years; (3) Multi-focal single system or multi-system involvement; (4) ECOG PS 0-2 score
  Interventions: Drug: Selinexor; Drug: Thalidomide (100mg); Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — The combined treatment period includes 12 cycles: receiving Selinexor (60mg, D1, 8, 15, 22), Thalidomide (100mg, D1-28), and Dexamethasone (40mg, D1, 8, 15, 22) as oral treatment, with each cycle lasting 28 days, for a total of 12 cycles of combined treatment, or until disease progression, death, or occurrence of intolerable toxicity. Alternatively, until disease progression, death, or occurrence of intolerable toxicity.
Drug: Thalidomide (100mg) — The combined treatment period includes 12 cycles: receiving Selinexor (60mg, D1, 8, 15, 22), Thalidomide (100mg, D1-28), and Dexamethasone (40mg, D1, 8, 15, 22) as oral treatment, with each cycle lasting 28 days, for a total of 12 cycles of combined treatment, or until disease progression, death, or occurrence of intolerable toxicity. Alternatively, until disease progression, death, or occurrence of intolerable toxicity.
Drug: Dexamethasone — The combined treatment period includes 12 cycles: receiving Selinexor (60mg, D1, 8, 15, 22), Thalidomide (100mg, D1-28), and Dexamethasone (40mg, D1, 8, 15, 22) as oral treatment, with each cycle lasting 28 days, for a total of 12 cycles of combined treatment, or until disease progression, death, or occurrence of intolerable toxicity. Alternatively, until disease progression, death, or occurrence of intolerable toxicity.

SUMMARY:
In adult patients with relapsed/refractory Langerhans cell histiocytosis (LCH), a treatment regimen of XTD regimen (Selinexor, Thalidomide and Dexamethasone) is planned to be used.

ELIGIBILITY:
Inclusion Criteria:

* Organ pathology confirmed diagnosis of LCH;
* Age 18 years or older;
* Multi-system involvement, or single system with multiple lesions;
* Disease not relieved after receiving at least one systemic treatment, or disease relapsed after improvement;
* ECOG performance status score ≤2;
* Clinical physician determines suitability for this treatment protocol;
* Subjects can understand the study protocol and are willing to participate in this study, providing written informed consent.

Exclusion Criteria:

* Single system single lesion LCH
* Underwent major surgery within 4 weeks prior to the first administration of the study drug;
* Underwent radiotherapy within 4 weeks prior to the first administration of the study drug;
* History of myocardial infarction within the past year; suffers from New York Heart Association (NYHA) class 3 or 4 congestive heart failure, or has a history of NYHA class 3 or 4 congestive heart failure, unless left ventricular ejection fraction (LVEF) ≥ 50% in the echocardiogram (ECHO) screening performed within 1 month before entering the study;
* Pregnant or breastfeeding women (women of childbearing age with positive pregnancy test at baseline or who have not undergone pregnancy testing. Postmenopausal women must have been menopausal for at least 12 months);
* Abnormal liver and kidney function: creatinine level ≥176.8μmol/l (2mg/dl), transaminase and bilirubin levels more than 2 times the upper limit of normal (for LCH patients with liver involvement, transaminase levels more than 10 times and bilirubin levels more than 3 times the upper limit of normal);
* Severe hematological abnormalities: absolute neutrophil count less than 1 × 10^9/L, platelet less than 50×10^9/L;
* Presence of uncontrolled infections;
* Any other circumstances that the investigator believes to be inappropriate for the patient to participate in this trial;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
PFS | From enrollment to the end of treatment at 8 weeks
  PFS defined as the time from XTD initiation to first documented disease progression, relapse after XTD, death from any cause, or last follow-up.

SECONDARY OUTCOMES:
ORR | From enrollment to the end of treatment at 8 weeks
  The overall response rate (ORR) was defined as the cumulative proportion of patients attaining either a complete response (CR) or partial response (PR) .
OS | From enrollment to the end of treatment at 8 weeks
  OS was measured from XTD initiation to death or last follow-up
Adverse Events | From enrollment to the end of treatment at 8 weeks
  Toxicities were recorded and graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

OTHER OUTCOMES:
Correlation between the positivity of NGS in MAPK pathway and therapeutic efficacy/PFS | From enrollment to the end of treatment at 8 weeks
  Correlation between the positivity of NGS in MAPK pathway and therapeutic efficacy/PFS
Fact-G | From enrollment to the end of treatment at 8 weeks
  The score of Functional Assessment of Cancer Therapy - General

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, beijing,, Beijing, China

IPD SHARING:
Plan to Share IPD: No